CLINICAL TRIAL: NCT01290458
Title: The Effect of Antioxidant Vitamin Supplementation on Muscle Performance and Redox Status After Eccentric Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: European University Cyprus (Other); Greek Ministry of Development (Other Government); Democritus University of Thrace (Other)
Responsible Party: Athanasios Jamurtas Dr, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: UTH-2008
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-01

CONDITIONS: Muscle Damage; Oxidative Stress; Hemolysis
Keywords: Eccentric training; Free radicals; Antioxidant supplements; Training adaptations; Lipid profile
MeSH Terms: conditions — Hemolysis | interventions — Ascorbic Acid; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin (Experimental)
  Interventions: Dietary Supplement: Antioxidant vitamins
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Antioxidant vitamins

INTERVENTIONS:
Dietary Supplement: Antioxidant vitamins — Oral supplementation with one tablet of 1 g of vitamin C (Lamberts Healthcare Ltd, UK) and one tablet of 400 IU of vitamin E (Lamberts Healthcare Ltd, UK)
  Other Names: For vitamin C ascorbic acid; For vitamin E d-alpha tocopherol

SUMMARY:
Consumption of vitamin supplements is a common practice among athletes or people participating in health promoting exercise programs. The reason for this interest in vitamin supplements is primarily because of the observation that enhanced production of reactive oxygen and nitrogen species (RONS) influence fundamental biological processes, such as gene expression, signal transduction and enzyme activity. In a muscle and exercise physiology context, a low level of RONS is required for normal force production, whereas marked increases in RONS can cause contractile dysfunction, resulting in muscle weakness and fatigue. On the other hand RONS are involved in signaling pathways and serve to up-regulate the expression of a number of genes and can exert favorable effects such as training adaptations.

The present study will employ a valid eccentric exercise model to examine the influence of combined vitamin C and E supplementation after acute and chronic eccentric exercise on muscle damage and performance, redox status, hemolysis and lipid and lipoprotein profile.

DETAILED DESCRIPTION:
Historically there was a shift in the paradigm regarding the effects of antioxidant supplementation on muscle performance and redox status. In fact, back in the 80's and 90's most of the relevant studies reported "positive" effects of antioxidant supplementation on muscle performance, muscle damage and redox status. On the other hand, the last five years, an increasing number of well-received studies are appearing pointing towards the negative impact of antioxidant supplementation. Moreover, much more studies than the past are now specifically addressing the effects of antioxidant supplementation on the exercise adaptations that take place after chronic exercise. Regarding the latter, it has been reported recently that antioxidant supplementation greatly decreases training efficiency and prevents many cellular adaptations to chronic exercise. Nevertheless, the debate is still open and an equal number of recent studies have reported the reverse i.e. positive effects of antioxidant supplementation on exercise adaptations or virtually no effect of antioxidant supplementation on exercise adaptations.

Eccentric muscle work is an essential part of daily activities of humans, such as walking, and in particular, when walking downhill or descending stairs. The most notable and well-described effect of eccentric exercise is the muscle damage that peaks one to three days after exercise. Eccentric exercise can cause effects other than just muscle damage, from activation of several transcription factors to favorable changes on lipid and lipoproteins profile.

In a double-blinded fashion, men will receive either a daily oral supplementation of vitamin C (1g) and vitamin E (400IU) or placebo for eleven weeks. Following baseline tests, volunteers will have to perform an eccentric exercise session two times per week for four weeks. Before and after the chronic eccentric exercise volunteers will be subject to one session of acute eccentric exercise, and physiological measurements will be performed as well as blood samples and muscle biopsies will be collected.

The aims of the present research are to investigate:

* the effect of antioxidant vitamin supplementation for 4 weeks on muscle performance, redox status, hemolysis and lipids and lipoprotein profile,
* the effect of an acute bout of eccentric exercise on muscle performance, redox status, hemolysis and lipid and lipoproteins profile of untrained individuals supplemented with or without antioxidant vitamins,
* the effect of 4 weeks of eccentric training on muscle performance, redox status, hemolysis and lipid and lipoproteins profile of untrained individuals supplemented with or without antioxidant vitamins,
* the effect of an acute bout of eccentric exercise on muscle performance, redox status, hemolysis and lipid and lipoproteins profile of individuals trained for 4 weeks and supplemented with or without antioxidant vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Physiological body mass index (BMI)
* Physiological health profile
* Subject provides written informed consent

Exclusion Criteria:

* Smoker
* Professional athlete
* Consumed any nutritional supplement the last 3 months
* Performed pure eccentric exercise the last 6 months
* Non Caucasian

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum isometric torque (torque) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  An isokinetic dynamometer (Cybex, Ronkonkoma, NY) will be used for the measurement of isometric knee extensor peak torque at 90° knee flexion. The average of the three best maximal voluntary contractions with their dominant leg will be recorded. In order to ensure that the subjects provide their maximal effort, the measurements will be repeated if the difference between the lower and the higher torque value exceeded 10%. There will be two minutes rest between isometric efforts.
Range of motion, ROM (degrees) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  The assessment of pain-free ROM will be performed manually using the the isokinetic dynamometer. The investigator will move the calf at a very low angular velocity from 0 knee extension to the position where the subject will feel any discomfort.
Delayed onset muscle soreness, DOMS (scale 1-10) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Each participant will assess delayed onset muscle soreness (DOMS) during squat movement (90o knee flexion) and perceived soreness will be rated on a scale ranging from 1 (normal) to 10 (very sore).
Creatine kinase, CK (activity IU) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  CK activity will be measured as a general indicator of muscle damage.It will be measured in a Cobas Integra Plus 400 chemistry analyzer. CK will be measured before the beginning of the supplementation (week 0), before and the week after the first bout of eccentric exercise (week 5), before and the week after the second bout of eccentric exercise (week 11).

SECONDARY OUTCOMES:
Reduced glutathione, GSH (μmol/g Hb) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  GSH will be measured as a general index of oxidative stress. For GSH, 20 μL of erythrocyte lysate will be treated with 5% TCA mixed with 660 μL of 67 mM sodium potassium phosphate (pH 8.0) and 330 ΜL of 1 mM 5,5-dithiobis-2 nitrobenzoate. The samples will be incubated in the dark at room temperature for 45 min, and the absorbance will be read at 412 nm.
Oxidized glutathione, GSSG (μmol/g Hb) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  GSSG will be measured as a general index of oxidative stress. It will be assayed by treating 50 μL of erythrocyte lysate with 5% TCA and neutralized up to pH 7.0-7.5. One microliter of 2-vinylpyridine will be added, and the samples will be incubated for 2 h. Sample will be treated with TCA and will be mixed with 600 μL of 143 mM sodium phosphate 100 ΜL of 3 mM NADPH, 100 ΜL of 10 mM 5,5-dithiobis-2-nitrobenzoate, and 194 μL of distilled water. After the addition of 1 μL of glutathione reductase, the change in absorbance at 412 nm will be read for 3 min.
Thiobarbituric acid-reactive substances, TBARS (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  TBARS will be measured as an index of lipid peroxidation. For TBARS determination, 100 μL of plasma will be mixed with 500 ΜL of 35% TCA and 500 μL of Tris-HCl (200 mM, pH 7.4) and will be incubated for 10 min at room temperature. One milliliter of 2 M Na2SO4 and 55 mM thiobarbituric acid solution will be added, and the samples will be incubated at 95 C for 45 min. The samples will be cooled on ice for 5 min and then will be vortexed after adding 1 mL of 70% TCA. The samples will be centrifuged at 15,000g for 3 min, and the absorbance of the supernatant will be read at 530 nm.
Protein carbonyls (nmol/mg pr.) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Carbonyls will be measured as an index of protein oxidation. Protein carbonyls will be determined adding 50 μL of 20% TCA to 50 μL of plasma. Samples will be incubated in the dark at room temperature for 1 h. The supernatant will be discarded, and 1 mL of 10% TCA will be added. The supernatant will be discarded, and 1 mL of ethanol-ethyl acetate will be added and centrifuged. The supernatant will be discarded, and 1 mL of 5 M urea will be added, vortexed, and incubated at 37C for 15 min. The samples will be centrifuged at 15,000g for 3 min at 4C, and the absorbance will be read at 375 nm.
Catalase (μmol/min/mg Hb) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Catalase will be measured as one of the main antioxidant enzyme of erythrocytes. Catalase activity will be determined adding 4 μL of erythrocyte lysate, 2955 μL of 67 mM sodium potassium phosphate (pH 7.4), and the samples will be incubated at 37C for 10 min. Five microliters of 30% hydrogen peroxide was added to the samples, and the change in absorbance will immediately read at 240 nm for 1.5 min.
Total antioxidant capacity, TAC (mm DPPH) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  TAC will be determined adding 20 μL of plasma to 480 ΜL of 10 mM sodium potassium phosphate (pH 7.4) and 500 μL of 0.1 mM 2,2-diphenyl-1-picrylhydrazyl (DPPH) free radical, and the samples will be incubated in the dark for 30 min at room temperature. The samples will be centrifuged for 3 min at 20,000g, and the absorbance will be read at 520 nm.
Albumin (g/L) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Albumin will be measured as an antioxidant component of blood plasma. It will be determined spectrophotometrically based on the formation of a coloured complex with bromocresol green reagent.
Uric acid (μm) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Uric acid will be measured as the main antioxidant component of blood plasma. It will be measured in a Cobas Integra Plus 400 chemistry analyzer.
Vitamin C and E (mmol/L) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Vitamin C will be measured in plasma using a ferric reducing ascorbate assay kit using spectrophotometry. Vitamin E will be measured in plasma with the use of HPLC.
Plasma hemoglobin (g/dL) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Plasma hemoglobin will be assayed with a commercial kit using spectrophotometry as a hemolysis index.
Bilirubin (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  Bilirubin will be measured in a Cobas Integra Plus 400 chemistry analyzer as a hemolysis index.
Triacylglycerols, TG (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  TG will be measured in a Cobas Integra Plus 400 chemistry analyzer.
Total cholesterol (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  TC will be measured in a Cobas Integra Plus 400 chemistry analyzer.
High-density lipoprotein cholesterol, HDLC (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  HDLC will be measured in a Cobas Integra Plus 400 chemistry analyzer.
Low-density lipoprotein cholesterol, LDLC (μM) | Before the beginning of the supplementation (week 0), the week after the first bout of eccentric exercise (week 5), and the week after the second bout of eccentric exercise (week 11)
  LDLC will be measured in a Cobas Integra Plus 400 chemistry analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, Dr, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Trikala, Greece

REFERENCES:
- [Background] Paschalis V, Nikolaidis MG, Theodorou AA, Panayiotou G, Fatouros IG, Koutedakis Y, Jamurtas AZ. A weekly bout of eccentric exercise is sufficient to induce health-promoting effects. Med Sci Sports Exerc. 2011 Jan;43(1):64-73. doi: 10.1249/MSS.0b013e3181e91d90. PMID 20508540
- [Background] Paschalis V, Nikolaidis MG, Giakas G, Theodorou AA, Sakellariou GK, Fatouros IG, Koutedakis Y, Jamurtas AZ. Beneficial changes in energy expenditure and lipid profile after eccentric exercise in overweight and lean women. Scand J Med Sci Sports. 2010 Feb;20(1):e103-11. doi: 10.1111/j.1600-0838.2009.00920.x. Epub 2009 Apr 14. PMID 19422638
- [Background] Nikolaidis MG, Paschalis V, Giakas G, Fatouros IG, Sakellariou GK, Theodorou AA, Koutedakis Y, Jamurtas AZ. Favorable and prolonged changes in blood lipid profile after muscle-damaging exercise. Med Sci Sports Exerc. 2008 Aug;40(8):1483-9. doi: 10.1249/MSS.0b013e31817356f2. PMID 18614942